CLINICAL TRIAL: NCT03253224
Title: The Influence of Intraoperative Magnesium Sulfate Administration on Postoperative Pain After Total Knee Arthroplasty in Patients Sedated With Dexmedetomidine Under Spinal Anesthesia: A Randomized-controlled Trial
Brief Title: Magnesium and Postoperative Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Because the principle investigator will participate a visiting scholar program for one year in other country, this study has been terminated.
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Jung Shin, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: B-1707/406-006
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2017-12

CONDITIONS: Arthritis Knee; Magnesium Sulfate; Dexmedetomidine
MeSH Terms: interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline (Placebo Comparator): Patient who received normal saline during the operation
  Interventions: Drug: Normal saline
- Magnesium (Experimental): Patient who received magnesium sulfate during the operation
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Magnesium group receives magnesium sulfate (50 mg/kg) in 100 mL of normal saline over 15 min during induction of anesthesia, followed by a continuous magnesium sulfate infusion (15 mg/kg/h) until the end of surgery.
  Arms: Magnesium
Drug: Normal saline — Normal saline group receives the same volume of normal saline, administered according to the same method as in the magnesium group.
  Arms: Saline

SUMMARY:
With ongoing advancements in healthcare leading to prolonged life expectancy, orthopedic surgeries are increasingly performed in elderly patients. Total knee arthroplasty, in particular, has been increasing with the growing demand for improved mobility and quality of life. Total knee arthroplasty is performed on patients with advanced and painful osteoarthritis of the knees, but it can result in moderate to severe postoperative pain during the recovery period.

To relieve anxiety or stress during surgery under regional anesthesia, sedation can be provided. Dexmedetomidine is a sedative-analgesic agent acting as α2-adrenergic receptor agonist, and its analgesic effect has been well established in various procedures or surgeries.

Magnesium has been reported to produce important analgesic effects including the suppression of neuropathic pain, potentiation of morphine analgesia, and attenuation of morphine tolerance. Although the exact mechanism is not yet fully understood, the analgesic properties of magnesium are believed to stem from regulation of calcium influx into the cell and antagonism of N-methyl-D-aspartate (NMDA) receptors in the central nervous system. In this study, investigators will evaluate the reducing effect of magnesium on the post-total knee arthroplasty pain in patients sedated with dexmedetomidine under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo total knee arthroplasty under spinal anesthesia
* Patients who want to sedation during the surgery
* American Society of Anesthesiologists physical status classification 1 and 2

Exclusion Criteria:

* General anesthesia
* Patients who do not want to sedation during the surgery
* Patients who do not receive patient controlled analgesia postoperatively
* Muscular disease
* Hypermagnesemia
* Atrioventricular block

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Patient controlled analgesia (PCA) | Postoperative 24 hour
  Amounts of PCA consumption

SECONDARY OUTCOMES:
Numerical rating scale | Postoperative 24 hour
  Postoperative pain score
Rescue analgesics | Postoperative 24 hour
  Amounts of the analgesics administered to mange the postoperative pain
Nausea | Postoperative 24 hour
  Incidence of nausea
Vomiting | Postoperative 24 hour
  Incidence of vomiting
Antiemetics | Postoperative 24 hour
  Amounts of antiemetics consumption

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Jung Shin, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No